CLINICAL TRIAL: NCT01424540
Title: A Randomized, Double Blind, Single Dose, Cross-Over Study to Assess the Cardiovascular Effects of GSK2336805 in Healthy Adult Volunteers
Brief Title: Cross-Over Study to Assess the Cardiovascular Effects of GSK2336805
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 115535
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — GSK2336805

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): GSK2336805 150mg
  Interventions: Drug: GSK2336805 150mg
- Treatment B (Placebo Comparator): GSK2336805 Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK2336805 150mg — Single Dose
  Arms: Treatment A
Other: Placebo — Single Dose
  Arms: Treatment B

SUMMARY:
This is a single-center, randomized, two part, double-blind, crossover study in healthy adult subjects to assess the effect of a single dose of GSK2336805 150mg on cardiac function comparing with placebo using echocardiography as a primary assessment modality

ELIGIBILITY:
Inclusion Criteria:

* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin less than or equal to 1.5xUpper Limit of Normal (ULN).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including [medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included at the discretion of the Investigator only if the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, oophorectomy, or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea.

Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the follow up visit.

* Body weight greater than or equal to 50 kilogram (kg) for men and 45 kg for women. Body mass index (BMI) between 18.5-30 inclusive will be allowed.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subject has demonstrated an adequate echocardiographic window.
* QTcB less than 450 milliseconds (msec).

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen,positive Hepatitis C antibody, or a positive test for HIV antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* History of regular alcohol consumption within 6 months of the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mililiters within a 56 day period.
* Pregnant females as determined by positive [serum or urine] hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice [and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices] from 7 days prior to the first dose of study medication.
* Left ventricular ejection fraction less than 55% at screening.
* The subject's systolic blood pressure is outside the range of 90-140, or diastolic blood pressure is outside the range of 45-90 or heart rate is outside the range of 50-100beats per minute for female subjects or 45-100 beats per minute for male subjects.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination):

Males-Heart rate less than 45 and greater than 100 beats per minute (bpm). Females-Heart rate less than 50 and greater than 100 bpm Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).

Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome). Sinus Pauses greater than 3 seconds. Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject. Non-sustained or sustained ventricular tachycardia ( greater than or equal to 3 consecutive ventricular ectopic beats).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2011-10-03 (Actual); Study Completion 2011-10-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with a change in ejection fraction greater than 10 percent | 10 hours
  Echocardiographic measures of contractility

SECONDARY OUTCOMES:
Number of subjects with electrocardiogram (ECG) parameters out of range | 3 hours
  Cardiovascular measures
Number of subjects with vital signs out of range | 24 hours
  Cardiovascular measures
Number of subjects with adverse events | 24 hours
  tolerability
Number of subjects using concurrent medication | 24 hours
  Concomitant medications
Number of subjects with laboratory values out of range | 24 hours
  Labs
Area under the curve (0-24) | 24 hours
  PK parameter
Maximum observed concentration (Cmax) | 24 hours
  PK parameter
Terminal phase half-life | 24 hours
  PK parameter
Lag time before observation of drug concentrations in sampled matrix | 24 hours
  PK parameter
Time of occurrence of Cmax | 24 hours
  PK parameter
Concentration at 24 hours | 24 hours
  PK parameter
Correlation between concentration and various safety parameters | 24 hours
  Safety, PK
B-type natriuretic peptide (BNP) lab result | 24 hours
  Cardiac biomarkers
Troponin lab results | 24 hours
  Cardiac biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Derived] Wilfret DA, Adkison KK, Jones LA, Lou Y, Gan J, Spreen W. Echocardiogram study to evaluate the effect of the novel hepatitis C virus NS5A inhibitor GSK2336805 on cardiac contractility in healthy subjects. Antimicrob Agents Chemother. 2013 Oct;57(10):5141-3. doi: 10.1128/AAC.00668-13. Epub 2013 Jul 15. PMID 23856771
- See also: Results for study 115535 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115535?search=study&study_ids=115535#rs